CLINICAL TRIAL: NCT05388331
Title: The Radiologically Isolated Syndrome International Cohort
Brief Title: RIS International Cohort
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 22Neuro01
Record Dates: First submitted 2022-04-19; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Multiple Sclerosis; Radiologically Isolated Syndrome
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, plasma, tears, CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- RIS/1-2 criteria
  Interventions: Other: No intervention
- RIS/3-4 criteria
  Interventions: Other: No intervention
- NON RIS/0 criteria
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The Radiologically Isolated Syndrome (RIS) corresponds to the discovery of white matter (WM) abnormalities suggestive of multiple sclerosis (MS) by their location, size, and appearance, on the brain or spinal cord Magnetic Resonance Imaging (MRI). This imaging is performed for a reason other than for suspicion of demyelinating disease in subjects without a history of neurological symptoms and a strict routine clinical neurological examination. It was defined and named in 2009 (Okuda et al.) after publishing 3 case series (French, USA, Turkey). The Radiologically Isolated Syndrome Consortium (RISC) published a cohort of subjects with an extended follow-up after the first brain MRI of MS, with 34% presenting an event (clinical conversion) at five years, 51.2 % of these subjects showed an event at ten years. The patients who offer a higher risk of developing a first clinical demyelinating event were identified such as male sex, young age, the presence of oligoclonal bands (BOCs) in the Cerebrospinal Fluid (CSF), the presence of infratentorial lesions and spinal cord lesions on the first MRI suggestive of RIS. The location and morphology of the lesions appear to be decisive for studying the risk of conversion. Our first objective is to prospectively collect data to identify the subjects who present a higher risk of developing a first clinical demyelinating event and the progression of the disease in these subjects.

Among the objectives of this worldwide cohort is the analysis of (1) environmental factors (Vit D, EBV, tobacco…), (2) MRI biomarkers, including atrophy, central veins signs, paramagnetic rings, and DTI.

(3) digital biomarkers (4) oculography (5) biological markers To summarize, this cohort will allow for analyzing features in imaging, biology and the exploration of digital and oculographic characteristics to identify predictive factors of clinical evolution of a large cohort of subjects presenting WM abnormalities suggestive of multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* white matter T2 lesions suggestive of demyelination
* asymptomatic
* normal neurological exam

Exclusion Criteria:

* abnormal neurological exam,
* suspicion of another disease explaining MRI lesions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects demonstrating white matter T2 lesion suggestive of demyelination, asymptomatic with a normal neurological exam, corresponding to RIS diagnostic criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-04-15 (Estimated); Study Completion 2029-04-15 (Estimated)

PRIMARY OUTCOMES:
Identification of lesions T2-weighted sequence at the index scan | at inclusion
  number of T2-weighted sequence
Identification of lesions T2-weighted sequence at the index scan | at inclusion
  localisation of interest of T2 lesion (juxtacortical, periventricular, infratentorial, spinal cord)
Identification of lesions T1 sequence with and without Gd at the index scan. | at inclusion
  Lesions number
Identification of lesions T1 sequence with and without Gd at the index scan. | at inclusion
  localisation of interest
Radiological progression : new T2 lesions | year 1
  localisation of interest
Radiological progression : new contrast enhancing lesions | year 1
  Lesions number
Radiological progression : new contrast enhancing lesions | year 1
  localisation of interest
Brain atrophy | year 1
  measurement of global and regional grey matter volume measurement of global and regional white matter volume
Brain atrophy | year 2
  measurement of global and regional grey matter volume measurement of global and regional white matter volume
Brain atrophy | year 3
  measurement of global and regional grey matter volume measurement of global and regional white matter volume
Brain atrophy | year 4
  measurement of global and regional grey matter volume measurement of global and regional white matter volume
Brain atrophy | year 5
  measurement of global and regional grey matter volume measurement of global and regional white matter volume
Brain atrophy | MS onset assessed up to 2 years
  measurement of global and regional grey matter volume measurement of global and regional white matter volume
Radiological progression : new T2 lesions | year 2
  number of T2-weighted sequence
Radiological progression : new T2 lesions | year 2
  localisation of interest of T2 lesion
Radiological progression : new T2 lesions | year 3
  number of T2-weighted sequence
Radiological progression : new T2 lesions | year 4
  localisation of interest of T2 lesion
Radiological progression : new T2 lesions | year 5
  number of T2-weighted sequence
Radiological progression : new T2 lesions | MS onset assessed up to 2 years
  localisation of interest of T2 lesion
Radiological progression : new contrast enhancing lesions | year 2
  localisation of interest
Radiological progression : new contrast enhancing lesions | year 2
  Lesions number
Radiological progression : new contrast enhancing lesions | year 3
  Lesions number
Radiological progression : new contrast enhancing lesions | year 3
  localisation of interest
Radiological progression : new contrast enhancing lesions | year 4
  Lesions number
Radiological progression : new contrast enhancing lesions | year 4
  localisation of interest
Radiological progression : new contrast enhancing lesions | year 5
  Lesions number
Radiological progression : new contrast enhancing lesions | year 5
  localisation of interest
Radiological progression : new contrast enhancing lesions | MS onset assessed up to 2 years
  Lesions number
Radiological progression : new contrast enhancing lesions | MS onset assessed up to 2 years
  localisation of interest

SECONDARY OUTCOMES:
Collect biological data | At inclusion
  number of plasma samples
Collect biological data | MS onset assessed up to 2 years
  number of plasma samples
Collect digital markers | at inclusion
  The number of abnormalities identified by the eVOG application correlated with cerebral atrophy
Collect digital markers | year 1
  Progression of the number of abnormalities identified by the eVOG application correlated with cerebral atrophy
Collect digital markers | year 2
  Progression of the number of abnormalities identified by the eVOG application correlated with cerebral atrophy
Collect digital markers | year 3
  Progression of the number of abnormalities identified by the eVOG application correlated with cerebral atrophy
Collect digital markers | year 4
  Progression of the number of abnormalities identified by the eVOG application correlated with cerebral atrophy
Collect digital markers | year 5
  Progression of the number of abnormalities identified by the eVOG application correlated with cerebral atrophy
Collect digital markers | MS onset assessed up to 2 years
  Progression of the number of abnormalities identified by the eVOG application correlated with cerebral atrophy

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No